CLINICAL TRIAL: NCT03020017
Title: A Phase 0 First-In-Human Study Using NU-0129: A Spherical Nucleic Acid (SNA) Gold Nanoparticle Targeting BCL2L12 in Recurrent Glioblastoma Multiforme or Gliosarcoma Patients
Brief Title: NU-0129 in Treating Patients With Recurrent Glioblastoma or Gliosarcoma Undergoing Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Priya Kumthekar, Priya Kumthekar, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16C01; STU00203790 (CTRP (Clinical Trial Reporting Program)); NU 16C01 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-02007 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Gliosarcoma; Recurrent Glioblastoma
MeSH Terms: conditions — Gliosarcoma; Glioblastoma | interventions — Molecular Targeted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NU-0129) (Experimental): Patients receive NU-0129 IV over 20-50 minutes and undergo standard of care tumor resection within 8-48 hours.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Targeted Molecular Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Targeted Molecular Therapy — Given NU-0129 IV
  Other Names: molecularly targeted therapy

SUMMARY:
The purpose of this research study is to evaluate the safety of the study drug, NU-0129, based on Spherical Nucleic Acid (SNA) platform when infused in patients with recurrent glioblastoma multiforme or gliosarcoma. The SNA consists of nucleic acids arranged on the surface of a small spherical gold nanoparticle. This is a first-in-human trial to determine the safety of NU-0129. NU-0129 can cross the blood brain barrier (a filtering mechanism that carry blood to the brain). Once within the tumor, the nucleic acid component is able to target a gene called Bcl2L12 that is present in glioblastoma multiforme, and is associated with tumor growth. This gene prevents tumor cells from apoptosis, which is the process of programmed cell death, thus promoting tumor growth. Researchers think that targeting the Bcl2L12 gene with NU-0129 will help stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of intravenous NU-0129 in patients with recurrent glioblastoma multiforme (GBM) or gliosarcoma (GS).

SECONDARY OBJECTIVES:

I. To analyze drug concentration in serum at specific time points after drug administration.

II. To demonstrate intratumoral penetration of NU-0129. III. To assess the feasibility of giving NU-0129 as a standard treatment for recurrent GBM or GS.

TERTIARY OBJECTIVES:

I. To analyze tumor tissue for Bcl2L12 expression levels after NU-0129 administration.

II. Preliminary response (progression free survival [PFS] and overall survival [OS] at 6 months; overall response rate [ORR]).

OUTLINE:

Patients receive NU-0129 intravenously (IV) over 20-50 minutes and undergo standard of care tumor resection within 8-48 hours.

After completion of study treatment, patients are followed up at 7, 14, 21, and 28 days and then every 84 days for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven glioblastoma multiforme (GBM) or gliosarcoma (GS)
* Patients must have measurable disease by Response Assessment in Neuro-Oncology (RANO) 2010 criteria at the time of registration (pre-operative)
* Patients must have failed at least one regimen of chemo or radiation therapy; NOTE: There is no limit to the number or types of prior therapy
* The patient must be a candidate for surgical debulking (either subtotal or gross total resection); biopsy-only candidates will not be eligible
* All patients must be capable to voluntarily sign an informed consent indicating that they are aware of the investigational nature of this study prior to registration
* Patients must have a Karnofsky performance status of >= 70
* Patients must have adequate bone marrow, liver, coagulation and renal function within 7days prior to study registration, as defined below:
* White blood cell count (WBC) >= 3,000/uL
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3 (Note: Transfusion or growth factor may be used for eligibility outside of 7 days)
* Hemoglobin >= 8 mg/dL (Note: Transfusion may be used for eligibility outside of 7 days)
* Bilirubin =< 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2 x ULN
* Creatinine =< 1.5 x ULN
* Urine protein =< 3 x ULN
* Cholesterol =< 300 mg/dL
* International normalized ration (INR) =< 1.5 x ULN
* Prothrombin time (PT)/partial thromboplastin time (PTT) =< 1.5 x ULN
* Any patient who has had a recent surgery should have recovered from all effects of the surgery and be cleared by their surgeon
* Patients must have confirmed availability of archival or freshly biopsied tumor tissue meeting protocol-defined specifications (10 unstained slides) prior to study enrollment
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception (e.g. hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 28 days following completion of therapy; should a female patient, or a male patient's partner, become pregnant or suspect she is pregnant while participating in this study, the patient should inform her or his treating physician immediately

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test (either urine or serum) within 14 days prior to registration

Exclusion Criteria:

* Patients must not have any significant infections or medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate NU-0129
* Patients must not have a history of any other cancer unless they are in complete remission and off of all therapy for that disease for a minimum of 3 years

  * Note: Non-melanoma skin cancer or carcinoma in-situ of the cervix are exceptions and may be permitted after discussion with study quality assurance manager (QAM)
* Patients must not have had radiation therapy within 12 weeks prior to registration
* Patients must not have had prior cancer therapy (including biologic, cytotoxic, and experimental therapies, nitrosoureas, and Gliadel wafers or other surgically implantable antitumor treatment) within 21 days of registration; if questions arise, please ask the principal investigator (PI)

  * NOTE: Patients must not have Novocure within 24 hours
* Hormonal tumor therapies should not be administered within 14 days of registration; exceptions may be discussed with the PI
* Patients must not have symptomatic hypertension
* Patients with known human immunodeficiency virus (HIV) infection or chronic or acute hepatitis B or C are not eligible; Note: Patients do not need to have HIV, hepatitis B, or hepatitis C testing at screening
* Female patients who are pregnant or breast feeding are not eligible
* Patients are not eligible if they are unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kumthekar, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NU-0129 Treatment: NU-0129 will be administered inpatient at ~ 0.04mg/kg IV 8-48 hours once prior to scheduled tumor resection. Dose corresponds to 1/50th of the no-observed-adverse-event level.
Period: NU-0129
Arm/Group | NU-0129 Treatment
Started | 8
Completed | 8
Not Completed | 0
Period: Standard of Care Resection
Arm/Group | NU-0129 Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NU-0129 Treatment
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 55.5 [28 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: To evaluate the safety of intravenous NU-0129 in patients with recurrent GBM or GS, the number of adverse events will be assessed and will be graded according to the NCI's Common Terminology Criteria in Adverse Events (CTCAE) version 4.03 where the grading is as follows:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-threatening Grade 5: Fatal
Time Frame: Up to 21 days after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | NU-0129 Treatment
Number analyzed (Participants) | 8
Participants
  Experienced any AE | 8
  Experienced an AE related to NU-01289 | 4
  Experienced any SAE | 1
  Experienced an SAE related to NU-0129 | 0

2. Secondary Outcome: NU-0129 Concentration in Blood After Drug Administration Using Maximum Concentration
Description: Blood samples will be collected post-infusion to analyze drug concentration at specific time points after drug administration. Median plasma concentrations of NU-0129 were derived from time profiles for both Seven different small interfering RNA (siRNA) and gold (Au) concentrations, with Au plasma concentration determined by inductively coupled plasma mass spectrometry (ICP-MS) and siRNA concentration assessed by liquid chromatography-high performance liquid chromatography (LC-HPLC) using an atto dye-labeled PNA probe.
Time Frame: At 1, 3, 5, 10, 30, and 60 minutes, and 4, 8, and 24 hours post infusion
Measure: Median (95% Confidence Interval); unit: ng/ml
Arm/Group | NU-0129 Treatment
Number analyzed (Participants) | 8
ng/ml
  siRNA maximum observed plasma concentration | 62.1 [22.8 to 123]
  Au maximum observed plasma concentration | 4290 [3120 to 7140]

3. Secondary Outcome: Biodistribution of NU-0129 in Tumor Tissue
Description: Tissue will be collected during the scheduled surgery and assayed with Inductively Coupled Plasma Mass Spectrometry (ICP-MS) to analyze the concentration of particles in various parts of tumor tissue. To analyze spatial distribution of Au within tumor tissue, synchrotron XFM elemental maps of GBM tissue slices were acquired at micron and submicron resolution and matched to adjacent hematoxylin and eosin (H&E)- and Ki67-stained tumor sections. Approximate percentage of gold (Au) found in cancer cells is reported below.
Time Frame: At time of surgery
Population: 2 patients tumor resections resulted in insufficient amount of viable tumor tissue for ICP-MS analysis and were not included in this analysis
Measure: Median (Standard Deviation); unit: percentage of gold "Au"
Arm/Group | NU-0129 Treatment
Number analyzed (Participants) | 6
percentage of gold "Au" | 20.5 (8.15)

4. Secondary Outcome: Feasibility of Giving NU-0129 as a Standard Treatment
Description: Feasibility will be calculated as the rate of successful production, delivery, and administration of the investigational product and subsequent resection.
Time Frame: At time of infusion (8-48 hours prior to resection) and during surgery
Population: Patients who had drug infused and underwent subsequent resection
Measure: Count of Participants; unit: Participants
Arm/Group | NU-0129 Treatment
Number analyzed (Participants) | 8
Participants
  Number of patients who had drug infused successfully | 8
  Number of patient who underwent subsequent resection | 8

5. Secondary Outcome: NU-0129 Concentration in Blood After Drug Administration Using Half-life
Description: as for outcome 2
Time Frame: At 1, 3, 5, 10, 30, and 60 minutes, and 4, 8, and 24 hours post infusion
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | NU-0129 Treatment
Number analyzed (Participants) | 8
hours
  siRNA half-life | 0.06 [0.02 to 0.16]
  Au half-life | 18 [12 to 23]

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events from the time of NU-0129 infusion through 21 days post infusion
Arm/Group | NU-0129 Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NU-0129 Treatment (N=8)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NU-0129 Treatment (N=8)
Alkaline phosphatase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT03020017/Prot_SAP_000.pdf